CLINICAL TRIAL: NCT01613456
Title: Effect of S.Cerevisiae vs Placebo on the Improvement of Gastrointestinal Disorders,Especially During Irritable Bowel Syndrome. Randomized, Double-blind Study
Brief Title: Effect of Saccharomyces Cerevisiae on the Symptoms of Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lesaffre International (Industry)
Collaborators: BioFortis (Other); University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: PEC11010; ID RCB: 2011-A00915-36 (Other: French Health Products Safety Agency)
Record Dates: First submitted 2012-06-05; First posted 2012-06-07 (Estimated); Last update posted 2015-05-14 (Estimated); Status verified 2015-05

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Placebo (Placebo Comparator): Dicalcium phosphate, Maltodextrin and Magnesium stearate.
  Interventions: Dietary Supplement: Placebo
- Saccharomyces cerevisiae CNCM I-3856 (Experimental)
  Interventions: Dietary Supplement: Saccharomyces cerevisiae CNCM I-3856

INTERVENTIONS:
Dietary Supplement: Saccharomyces cerevisiae CNCM I-3856 — 2 capsules/day during 12 weeks
  Arms: Saccharomyces cerevisiae CNCM I-3856
Dietary Supplement: Placebo — Capsule with comparable organoleptic properties and weight than the experimental product.
  2 capsules/day during 12 weeks
  Arms: Placebo

SUMMARY:
The main purpose of this study is the effect of the probiotic yeast Saccharomyces cerevisiae CNCM I-3856 on abdominal pain or intestinal discomfort in patients presenting with the irritable bowel syndrome (IBS)

ELIGIBILITY:
Inclusion criteria:

* IBS subject meeting the Rome III criteria , with a discomfort or pain present more than 1 day per week in whom organic causes of their symptoms have been excluded
* IBS-C with less than 3 complete spontaneous bowel movements/week
* IBS-D with at least 2 or more days/week one stool which has consistency of type 6 or 7 Bristol stool score
* Subject able of and willing to comply with the protocol and to give their written informed consents

Exclusion criteria:

* History of chronic gastrointestinal disorders
* History of lactose intolerance
* History of gluten intolerance
* Treatment able to influence IBS, modifying intestinal sensitivity and motility (antidepressants,opioid, narcotic analgesics)
* Eating disorders
* Pregnancy in progress

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 364 (Actual)
Dates: Start 2011-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in discomfort score,obtained by Daily Likert Scale averaged by week | baseline and week 8

CONTACTS AND LOCATIONS:
Overall Officials: David GENDRE, MD, Principal Investigator — BioFortis; Robin SPILLER, Professor of Gastroenterology, Principal Investigator — Nottingham Digestive Diseases Centre University Hospital
Locations (1):
- Biofortis, Saint-Herblain, France

REFERENCES:
- [Derived] Spiller R, Pelerin F, Cayzeele Decherf A, Maudet C, Housez B, Cazaubiel M, Justen P. Randomized double blind placebo-controlled trial of Saccharomyces cerevisiae CNCM I-3856 in irritable bowel syndrome: improvement in abdominal pain and bloating in those with predominant constipation. United European Gastroenterol J. 2016 Jun;4(3):353-62. doi: 10.1177/2050640615602571. Epub 2015 Aug 21. PMID 27403301